CLINICAL TRIAL: NCT02752594
Title: Evaluation of the Consumption of Probiotics on the Bacteria Causing Dental Caries: A Randomised Clinical Trial
Brief Title: Consumption of Probiotics on Salivary Bacteria Causing Dental Caries
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sharda University (Other)
Responsible Party: Principal Investigator, G.RATNA VELUGU, Assistant Professor, Sharda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D22052015
Record Dates: First submitted 2016-04-18; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Dental Caries
Keywords: probiotic; mutans streptococci; bacillus coagulans; caries
MeSH Terms: conditions — Dental Caries | interventions — Probiotics; exopolysaccharide biopolymer, Bacillus coagulans

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- probiotic (Experimental): 2 mg of probiotic powder mixed in 10 ml of distilled water
  Interventions: Biological: probiotic; Other: placebo
- placebo (Placebo Comparator): 10 ml of distilled water
  Interventions: Biological: probiotic; Other: placebo

INTERVENTIONS:
Biological: probiotic — Probiotic was administered for a period of 14 consecutive days. Saliva was collected on Day 1, before intervention and on Day 15, after intervention
  Other Names: bacillus coagulans
Other: placebo — placebo was administered for a period of 14 consecutive days. Saliva was collected on Day 1, before intervention and on Day 15, after intervention

SUMMARY:
Dental caries is a multifactorial disease effecting majority of the human population.One of the etiological factor causing dental caries is salivary mutans streptococci. Reducing the levels of this bacteria in the saliva can significantly reduce the incidence of dental caries. A non-invasive intervention, such as the administration of probiotics reduced the salivary mutans streptococci levels.

DETAILED DESCRIPTION:
40 candidates were selected from a pre-determined group and were randomly assigned to two groups. Group A (n=20) was administered probiotic drink and Group B (n=20) was administered placebo for 14 consecutive days. Saliva was collected on day 1 and day 15 to compare the salivary mutans streptococci levels.

ELIGIBILITY:
Inclusion Criteria:

* Decayed Missing Filled Surfaces less than or equal to 6
* Brushes twice daily

Exclusion Criteria:

* undergoing orthodontic treatment
* topical fluoride therapy in the past 2 yrs
* using sugar free gums

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
counts of streptococcus mutans after the consumption of probiotic | 15 days
  Human saliva was assessed for the counts of streptococcus mutans, one of the major etiological factor for dental caries

CONTACTS AND LOCATIONS:
Overall Officials: G. RATNA VELUGU, MDS, Principal Investigator — Sharda University

IPD SHARING:
Plan to Share IPD: No